CLINICAL TRIAL: NCT04707170
Title: MRI Exploration of Meningeal Inflammatory Disease
Acronym: EIME
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2020_38
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI with gadolinium injection — Patients presenting for imaging for whom an MRI examination with gadolinium injection has been prescribed and who meet the inclusion and non-inclusion criteria will be offered to participate in the study.
  The patients included, hospitalized at the A. de Rothschild Foundation Hospital for at least 24 hours, may be included in the ancillary study to meet secondary objective number 5.

SUMMARY:
Patients who have agreed to participate in the study will complete the MRI protocol as part of routine care, to which two additional sequences of 6 minutes duration will be added.

The MRI of routine care includes at least the following sequences:

* 3D T1 TFE 1.0 isotropic (2 minutes)
* T2 TSE (2 minutes)
* 3D FLAIR pre-injection (opt) (3 minutes)
* 3D FLAIR post-injection (3 minutes)

As part of the research, the following sequences will be acquired:

* FABIR pre-injection (3 minutes)
* FABIR post-injection (3 minutes)

Patients hospitalized for a foreseeable duration of at least 24 hours will be offered participation in the longitudinal tab of the study, for which four non-injected MRI examinations will be performed. The examinations will be carried out remotely from the injected MRI (1h, 2h, 12h-15h, 24h-36h). These exams dedicated to research will include the following sequences for a maximum of 8 minutes:

* 3D T1 TFE 1.0 isotropic (2 minutes)
* 3D FLAIR (3 minutes)
* FABIR (3 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* To benefit as part of his treatment of an MRI with injection of gadolinium
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

For the ancillary study to meet secondary endpoint number 5:

* Patient over 18 years old
* To benefit as part of his treatment of an MRI with injection of gadolinium
* Hospitalized for an expected period of at least 48 hours after the time of inclusion
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for imaging for whom an MRI examination with gadolinium injection has been prescribed and who meet the inclusion and non-inclusion criteria will be offered to participate in the study.
  The patients included, hospitalized at the A. de Rothschild Foundation Hospital for at least 24 hours, may be included in the ancillary study to meet secondary objective number 5
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
detection of meningeal contrast enhancement with the flair sequence | 1 DAY
detection of meningeal contrast enhancement with the FABIR sequence | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: julien savatovsky, Principal Investigator — Hôpital fondation Adolphe de Rothschild
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No